CLINICAL TRIAL: NCT02569255
Title: Safe Use of New Oral Anticoagulants in Patients Treated by Catheter Ablation for Atrial Fibrillation
Brief Title: Safe Use of New Oral Anticoagulants in Ablation for Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Private Hospital Heart Center Varde (Other)
Responsible Party: Principal Investigator, Peter Steen Hansen, Chief Electrophysiologist, MD, Ph.D., DMSci, Private Hospital Heart Center Varde
Other Study IDs: NOAC and PVI 2015
Record Dates: First submitted 2015-10-01; First posted 2015-10-06 (Estimated); Last update posted 2015-10-06 (Estimated); Status verified 2015-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pulmonary venous ostia isolation — Percutaneous, catheterbased, radiofrequency ablation with left atrial access via atrial septal puncture. Helped by 3D-imaging system (Carto(tm)) and electrical signal guidance the PV ostia together with neighbouring atrial tissue is electrically isolated from the rest of the left atrium.
  Other Names: catheter ablation, PVI

SUMMARY:
Use of new oral anticoagulants (NOAC) in patients before and after catheter based pulmonary vein isolation (PVI) is still controversial. Experience is reported from consecutive patients ablated with PVI for atrial fibrillation and treated with dabigatran, rivaroxaban, or apixaban from Nov 2011 until Dec 2014. Patients are followed for 3 month after ablation. All complications possible being related to the use of NOAC are registered.

DETAILED DESCRIPTION:
Use of new oral anticoagulants (NOAC) in patients before and after radiofrequency ablation with pulmonary vein isolation (PVI) is still controversial. Experience is reported from consecutive patients ablated with PVI for atrial fibrillation and treated with dabigatran, rivaroxaban, or apixaban from Nov 2011 until Dec 2014. Patients paused their NOAC treatment for 24 hours before ablation. Patients were routinely followed up after 3 months with a standard formular focused on possible adverse events (major bleeding complications or thromboembolic events) to NOAC treatment. Adverse events related to the use of NOAC were registered during treatment or during 3 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic atrial fibrillation despite pharmacological treatment.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with paroxysmal or persistent atrial fibrillation and symptomatic despite pharmacological treatment.
Sampling Method: Non-Probability Sample
Enrollment: 234 (Actual)
Dates: Start 2011-11; Primary Completion 2014-12 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with bleeding or thromboembolism during PVI and/or three months of follow up | Up to three months after PVI
  Any bleeding or thromboembolism observed during the PVI procedure and/or during 3 months of follow-up are registered. Also, if any procedure related complication was worsened by treatment with NOAC was registered.

CONTACTS AND LOCATIONS:
Overall Officials: Peter S Hansen, M.D., Principal Investigator — Varde Heart Center